CLINICAL TRIAL: NCT07179640
Title: A Randomised, Placebo Controlled, Double-Blind, Single-Ascending Dose And Multiple-Ascending Dose First-In-Human Study To Investigate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Orally Administered ALE1 With Or Without Food In Healthy Adult Subjects And Adult Patients With Hypophosphatasia
Brief Title: A Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ALE1 in Healthy Adults and Adults With Hypophosphatasia in Order to Identify Suitable Doses of ALE1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alesta Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALE1-101
Record Dates: First submitted 2025-08-04; First posted 2025-09-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hypophosphatasia (HPP)
Keywords: hypophosphatasia
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1 Cohort A (Experimental)
  Interventions: Drug: ALE1; Drug: Placebo
- Part 1 Cohort B (Experimental)
  Interventions: Drug: ALE1; Drug: Placebo
- Part 2 Cohort A (Experimental)
  Interventions: Drug: ALE1; Drug: Placebo
- Part 2 Cohort B (Experimental)
  Interventions: Drug: ALE1; Drug: Placebo
- Part 1 Cohort C (Experimental)
  Interventions: Drug: ALE1; Drug: Placebo

INTERVENTIONS:
Drug: ALE1 — Specified dose on specified days
Drug: Placebo — Specified dose on specified days

SUMMARY:
This is a phase 1/2a randomised, placebo controlled, double-blind study investigating the safety, tolerability, pharmacokinetics, and pharmacodynamics of ALE1 on healthy adult subjects and adult patients with Hypophosphatasia (HPP).

ELIGIBILITY:
Key Inclusion Criteria Part 1:

1. Participants are overtly healthy as determined by a medical evaluation
2. No concurrent medical conditions or significant medical history, in the opinion of the investigator.

Key Inclusion Criteria Part 2:

1. Documented ALPL gene variant

Key Exclusion Criteria Part 1:

1. History of conditions affecting bone or mineral metabolism

Key Exclusion Criteria Part 2:

1. Previous treatment with an enzyme replacement therapy (ERT) or any advanced therapeutic agent (e.g., gene therapy) for the treatment of hypophosphatasia (HPP) or any treatment for osteoporotic diseases
2. Previous exposure to any medication or investigational agent potentially affecting bone structure, muscle volume, muscle strength, or muscle or nerve function
3. Diagnosis of hyperparathyroidism
4. Diagnosis of hypoparathyroidism, unless secondary to HPP
5. New fracture within 12 weeks before first dosing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of ALE1 by assessing the number of treatment emergent adverse events (TEAEs) | From baseline up to day 16
Evaluate safety of ALE1 by assessing the presence of clinically significant changes in participants haematology parameters post-dose | From baseline up to day 16
Evaluate safety of ALE1 by assessing the presence of clinically significant changes in participants biochemistry parameters post-dose | From baseline up to day 16
Evaluate safety of ALE1 by assessing changes in heart rhythms via electrocardiogram | From baseline up to day 16
Evaluate safety of ALE 1 by assessing the presence of clinically significiant changes in participants vital signs | From baseline up to day 16

SECONDARY OUTCOMES:
Pharmacokinetic parameter: area under the plasma concentration versus time curve (AUC (D0 - INF)) | From baseline up to day 16
Pharmacokinetic parameter: time at which maximum plasma concentration occurs (Tmax) | From baseline up to day 16
Pharmacokinetic parameter: terminal elimination phase half-life (t(1/2)) | From baseline up to day 16
Pharmacokinetic parameter: total clearance (CL/F) | From baseline up to day 16
Pharmacokinetic parameter: volume of distribution (Vd/F) | From baseline up to day 16
Change in pharmacodynamic biomarker levels in blood samples of ALE1 | From baseline up to day 16
Dose proportionality of maximum observed plasma concentration (Cmax) Time at which maximum plasma concentration occurs (Tmax) | From baseline up to day 16
Dose proportionality of area under the plasma concentration versus time curve (AUC (D0 - INF)) | From baseline up to day 16
Effect of food on area under the plasma concentration versus time curve (AUC (D0 - INF)) | From baseline up to 16 days post dose
Effect of food on maximum observed plasma concentration (Cmax) | From baseline up to day 16

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand Clinical Research, Grafton, Auckland, New Zealand
- Fortrea Clinical Research Unit, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No